CLINICAL TRIAL: NCT07185113
Title: A Phase 1, Single Dose, Open-label Study to Assess the Pharmacokinetics of GEn-1124 After Single Oral Dosing in Healthy Subjects
Brief Title: A Study to Assess the Pharmacokinetics of GEn-1124 After Single Oral Dosing in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GEn1E Lifesciences (Industry)
Collaborators: InClin, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEn-1124-003
Record Dates: First submitted 2025-08-11; First posted 2025-09-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult Male
Keywords: GEn-1124; Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single oral dose in healthy male volunteers (Experimental): There will be only one group of participants that will receive a single oral capsule dose, administered under fed conditions following a standardized meal.
  Interventions: Drug: GEn-1124

INTERVENTIONS:
Drug: GEn-1124 — GEn-1124 will be administered to one single dose group of subjects dosed under fed (standardized meal) conditions. GEn-1124 will be administered as an oral capsule formulation containing GEn-1124.

SUMMARY:
The goal of this clinical trial is to determine the pharmacokinetics (how the body interacts with administered substances for the entire duration of exposure) of Gen-1124 in an oral formulation (taken by mouth) in healthy volunteers. It will also learn about the safety of Gen-1124. The main questions it aims to answer are:

- How does Gen-1124 interact with a human body?

Researchers will look at how Gen-1124 interacts with the body and what side effects it may cause.

Participants will:

* Take Gen-1124 for a single dose
* Remain in clinic for 2 days for checkups and tests
* Recieve a phone call for a checkup 3 and 7 days after the single dose

DETAILED DESCRIPTION:
Approximately 6 healthy male subjects who meet all eligibility criteria will be dosed.

There will be one single dose group of subjects dosed under fed (standardized meal) conditions.

Screening will be initiated up to 28 days before dosing. A follow-up visit will be completed approximately 7 days after dosing. Thus, total duration of subject participation in the study, excluding the Screening visit, will be approximately 8 days.

The incidence of adverse events from the time of informed consent through the final follow-up visit (end of study). This will be based on the results of:

* Physical exams,
* Electrocardiography (ECG) results,
* Clinical laboratory results,
* Vital signs,
* Concomitant medications. Plasma levels of GEn-1124 and potential metabolites will be estimated using non-compartmental methods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects;
2. Between 18 and 55 years of age;
3. Provide a signed EC-approved consent form;
4. Generally healthy, in the opinion of the Investigator;
5. Body Mass Index (BMI) 18 to 32 kg/m^2;
6. Creatinine clearance with in specific parameter;
7. Using method of contraception;
8. Willing and able to comply with protocol requirements for the duration of the study.

Exclusion Criteria:

1. Subjects taking prohibited medication;
2. Subjects with a history or presence of clinically significant medical or psychiatric disease;
3. Subjects who have regularly used nicotine-containing products ;
4. Subjects who have used caffeine-containing products;
5. Subjects who are unable to comply with eating a standardized meal during the study;
6. Subjects with a hospital admission or major surgery within 30 days prior to Screening;
7. Subjects with a plasma donation within 7 days prior to Screening;
8. Subjects who have not abstained from alcoholic beverages/alcohol-containing products at least 72 hours prior to first dose, or plan to consume them at any time through completion of the Follow-up Visit;
9. Subjects who cannot refrain from strenuous exercise from 72 hours prior to dose administration through completion of the Follow-up Visit;
10. Subjects who have participated (taken investigative drug and/or device) in another clinical trial within 90 days prior to Screening;
11. Subjects who are employees of the study unit or their family members, students who are working in the study unit, or family members of the Investigator or Sponsor.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PK Endpoints - Plasma levels | From enrollment to Day 2 discharge
  Plasma levels of GEn-1124 and potential metabolites will be estimated using non-compartmental methods, including:
  • Peak concentration (Cmax)
PK Endpoints - Plasma levels | From enrollment to Day 2 discharge
  Plasma levels of GEn-1124 and potential metabolites will be estimated using non-compartmental methods, including:
  • Terminal elimination rate constant (Kel) and half-life (T1/2)
PK Endpoints - Plasma levels | From enrollment to Day 2 discharge
  Plasma levels of GEn-1124 and potential metabolites will be estimated using non-compartmental methods, including:
  • Area under the concentration-time curve (AUC)
PK Endpoints - Plasma levels | From enrollment to Day 2 discharge
  Plasma levels of GEn-1124 and potential metabolites will be estimated using non-compartmental methods, including:
  • Apparent Oral Clearance (CL/F)
PK Endpoints - Plasma levels | From enrollment to Day 2 discharge
  Plasma levels of GEn-1124 and potential metabolites will be estimated using non-compartmental methods, including:
  • Apparent Volume of distribution (V/F)
Safety Endpoints - Clinically significant changes to physical exam | From informed consent/screening visit to Day 2
  The incidence of adverse events related to changes to Complete Physical exam at screening and pre-dose. All other exams will be symptom-driven and performed at the very least on Day 2. Results will be reviewed for any abnormalities and clinical significance.
Safety Endpoints - Clinically significant changes to ECG results | From informed consent/screening visit to Day 2
  The incidence of adverse related to Electrocardiography (ECG) results, measured by the change from baseline ECG parameters at screening, pre-dose and Day 2. The following parameters will be reviewed: heart rate, QT interval, PR interval, QRS interval, and QT corrected interval (QTcF [Fredericia's]).
  All will be assessed as within normal limits, abnormal but not clinically significant, or abnormal and clinically significant on an ongoing basis. Comparison will be made by changes from baseline screening results.
Safety Endpoints - Clinically significant changes to clinical lab results | From informed consent/screening visit to Day 2
  The incidence of adverse events based on the results of Clinical laboratory results, measured at screening, pre-dose and Day 2. Clinical labs to include chemistry, haematology, coagulation, and urinalysis. Results will be reviewed for any abnormalities and clinical significance.
Safety Endpoints - Clinically significant changes to vital signs | From informed consent/screening visit to Day 2
  The incidence of adverse events based on the results of Vital signs, measured at screening, pre-dose and Day 2. This includes systolic/diastolic blood pressure (mmHg ), heart rate (beats per minute), temperature (◦C), and oxygen saturation (SpO2) via pulse oximetry). Results will be reviewed for any abnormalities and clinical significance.
Safety Endpoints - Changes to concomitant medications | From 14 days (or 5 half-lives, whichever is longer) prior to Screening through completion of the study.
  Changes in baseline concomitant medications recorded from 14 days (or 5 half-lives, whichever is longer) prior to Screening through completion of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research (NZCR), Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No